CLINICAL TRIAL: NCT03100058
Title: A Randomized, Double-blind, Dose-finding Study to Evaluate the Change in Weight After 24 Weeks Treatment With 8 Doses of LIK066 Compared to Placebo in Obese or Overweight Adults, Followed by 24 Weeks Treatment With 2 Doses of LIK066 and Placebo
Brief Title: A Study to Evaluate the Change in Weight After 24 Weeks Treatment With LIK066 in Obese or Overweight Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIK066B2201; 2016-002868-14 (EudraCT Number)
Record Dates: First submitted 2017-03-03; First posted 2017-04-04 (Actual); Results first posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — licogliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- LIK066 2.5mg qd (Epoch 3) (Experimental): LIK066 2.5mg qd (once daily) dosing frequency for 24 weeks.
  Interventions: Drug: LIK066
- Placebo (Epoch 3) (Placebo Comparator): Matching placebo tablets for 24 weeks
  Interventions: Drug: Placebo
- LIK066 10mg qd (Epoch 3) (Experimental): LIK066 10mg qd (once daily) dosing frequency for 24 weeks
  Interventions: Drug: LIK066
- LIK066 50mg qd (Epoch 3) (Experimental): LIK066 50mg qd (once daily) dosing frequency for 24 weeks
  Interventions: Drug: LIK066
- LIK066 150mg qd (Epoch 3) (Experimental): LIK066 150mg qd (once daily) dosing frequency for 24 weeks
  Interventions: Drug: LIK066
- LIK066 2.5mg bid (Epoch 3) (Experimental): LIK066 2.5mg bid (once daily) dosing frequency for 24 weeks
  Interventions: Drug: LIK066
- LIK066 5mg bid (Epoch 3) (Experimental): LIK066 5mg bid (once daily) dosing frequency for 24 weeks
  Interventions: Drug: LIK066
- LIK066 25mg bid (Epoch 3) (Experimental): LIK066 25mg bid (once daily) dosing frequency for 24 weeks
  Interventions: Drug: LIK066
- LIK066 50mg bid (Epoch 3) (Experimental): LIK066 50mg bid dosing frequency for 24 weeks
  Interventions: Drug: LIK066
- LIK066 qd/LIK066 25mg qd (Epoch 4) (Experimental): Between week 24 to week 48, the patients who received a once daily regimen in the first 24 weeks will receive Dose A of LIK066 once daily and patients who received a twice daily regimen in the first 24 weeks will receive Dose B LIK066 once daily
  Interventions: Drug: LIK066
- LIK066 bid/LIK066 35mg qd (Epoch 4) (Experimental): Between week 24 to week 48, the patients who received a once daily regimen in the first 24 weeks will receive Dose A of LIK066 once daily and patients who received a twice daily regimen in the first 24 weeks will receive Dose B LIK066 once daily
  Interventions: Drug: LIK066
- Placebo/LIK066 25mg qd (Epoch 4) (Experimental): Between week 24 to week 48, the patients who received a once daily regimen in the first 24 weeks will receive Dose A of LIK066 once daily and patients who received a twice daily regimen in the first 24 weeks will receive Dose B LIK066 once daily
  Interventions: Drug: LIK066
- Placebo/Placebo (Epoch 4) (Placebo Comparator): Between week 24 to week 48, the patients who received a once daily regimen in the first 24 weeks will receive Dose A of LIK066 once daily and patients who received a twice daily regimen in the first 24 weeks will receive Dose B LIK066 once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIK066 — LIK066 will be supplied in different doses as tablets to be taken orally.
  Arms: LIK066 10mg qd (Epoch 3); LIK066 150mg qd (Epoch 3); LIK066 2.5mg bid (Epoch 3); LIK066 2.5mg qd (Epoch 3); LIK066 25mg bid (Epoch 3); LIK066 50mg bid (Epoch 3); LIK066 50mg qd (Epoch 3); LIK066 5mg bid (Epoch 3); LIK066 bid/LIK066 35mg qd (Epoch 4); LIK066 qd/LIK066 25mg qd (Epoch 4); Placebo/LIK066 25mg qd (Epoch 4)
Drug: Placebo — Placebo
  Arms: Placebo (Epoch 3); Placebo/Placebo (Epoch 4)

SUMMARY:
This was a dose-finding study that evaluated the change in weight after 24 weeks treatment with 8 different doses of LIK066 compared to placebo in obese or overweight adults, followed by 24 weeks treatment with 2 doses of LIK066 and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. informed consent
2. (BMI>=30) or (BMI>=27 with history of CV disease, hypertension, dyslipidemia, pre-diabetes or type 2 diabetes mellitus, sleep-apnea syndrome)
3. willing to comply with life-style intervention and treatment during the full duration of the study (approximately 54 weeks)

Exclusion Criteria:

* Hypersensitivity to any of the study medications
* Pregnancy or lactating women
* History of malignancies
* Use of pharmacologically active weight loss products
* Bariatric surgery
* Ketoacidosis, lactic acidosis, hyperosmolar coma in the 6 months before the screening visit.
* HbA1c >10% at the screening visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2017-05-06 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (76):
- United States (55):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Jasper, Alabama
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Carmichael, California
  - Novartis Investigative Site, Concord, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Roseville, California
  - Novartis Investigative Site, San Ramon, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Golden, Colorado
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Athens, Georgia
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Gurnee, Illinois
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Wauconda, Illinois
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Covington, Louisiana
  - Novartis Investigative Site, Hammond, Louisiana
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Beltsville, Maryland
  - Novartis Investigative Site, Towson, Maryland
  - Novartis Investigative Site, Royal Oak, Michigan
  - Novartis Investigative Site, City of Saint Peters, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Hickory, North Carolina
  - Novartis Investigative Site, Lansdale, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Moncks Corner, South Carolina
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, Summerville, South Carolina
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Bountiful, Utah
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Newport News, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Renton, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Kenosha, Wisconsin
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Canada (3):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Lévis, Quebec
- Czechia (5):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, České Budějovice
  - Novartis Investigative Site, Olomouc Lazce
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Slaný
- Hungary (3):
  - Novartis Investigative Site, Csongrád
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Szentes
- Slovakia (3):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Sereď
- United Kingdom (5):
  - Novartis Investigative Site, Basingstoke
  - Novartis Investigative Site, Blackburn
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Rotherham
  - Novartis Investigative Site, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 674 patients were screened. Of the 460 patients who were randomized to the study, the majority (85.7%) completed Epoch 3. Of the 394 patients who completed Epoch 3 and entered Epoch 4, the majority (93.1%) completed the Epoch 4 study period.
Pre-assignment Details: Overall, 674 patients were screened. Of the 460 patients who were randomized to the study, the majority (85.7%) completed Epoch 3. Of the 394 patients who completed Epoch 3 and entered Epoch 4, the majority (93.1%) completed the Epoch 4 study period.
Groups:
- LIK066 2.5mg Bid (Epoch 3): LIK066 2.5mg bid (twice daily) dosing frequency for 24 weeks
- LIK066 5mg Bid (Epoch 3): LIK066 5mg bid (twice daily) dosing frequency for 24 weeks
- LIK066 25mg Bid (Epoch 3): LIK066 25mg bid (twice daily) dosing frequency for 24 weeks
- LIK066 50mg Bid (Epoch 3): LIK066 50mg bid (twice daily) dosing frequency for 24 weeks
- LIK066 qd/LIK066 25 mg qd (Epoch 4): LIK066 qd (once daily) patients who entered Epoch 4 and received LIK066 25 mg qd
- LIK066 Bid/LIK066 35 mg qd (Epoch 4): LIK066 bid patients who entered Epoch 4 and received LIK066 35 mg qd
- Placebo/LIK066 25 mg qd (Epoch 4): Matching placebo tablets for 24 weeks
- Placebo qd (Epoch 4): Placebo patients who entered Epoch 4 and received matching Placebo tablets qd
Period: Epoch 3 (24 Weeks of Treatment)
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3) | LIK066 qd/LIK066 25 mg qd (Epoch 4) | LIK066 Bid/LIK066 35 mg qd (Epoch 4) | Placebo/LIK066 25 mg qd (Epoch 4) | Placebo qd (Epoch 4)
Started | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78 | 0 | 0 | 0 | 0
Completed | 35 | 31 | 29 | 63 | 36 | 37 | 30 | 60 | 73 | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 9 | 14 | 2 | 2 | 8 | 16 | 5 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 4 | 8 | 1 | 0 | 3 | 11 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 3 | 4 | 1 | 1 | 1 | 4 | 2 | 0 | 0 | 0 | 0
Not completed — Non-compliance with study treatment | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Epoch 4 (Last 24 Weeks of the Study)
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3) | LIK066 qd/LIK066 25 mg qd (Epoch 4) | LIK066 Bid/LIK066 35 mg qd (Epoch 4) | Placebo/LIK066 25 mg qd (Epoch 4) | Placebo qd (Epoch 4)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 158 | 163 | 39 | 34
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 153 | 148 | 36 | 30
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 15 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — non-compliance with study treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3) | Total
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78 | 460
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (12.20) | 53.2 (10.08) | 52.9 (13.60) | 51.1 (12.94) | 53.4 (12.28) | 49.8 (11.50) | 49.7 (11.93) | 52.9 (11.87) | 51.1 (13.27) | 51.7 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 25 | 44 | 20 | 24 | 26 | 49 | 45 | 283
  Male | 15 | 11 | 13 | 33 | 18 | 15 | 12 | 27 | 33 | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 6
  Asian | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 5 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3
  Black or African American | 5 | 4 | 5 | 5 | 2 | 3 | 4 | 6 | 8 | 42
  White | 30 | 33 | 33 | 67 | 36 | 32 | 34 | 63 | 64 | 392
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight at 24 Weeks
Description: Dose-response relationship of two dose regimens of LIK066 as measured by the percent change from baseline in body weight relative to placebo after 24 weeks of treatment
Time Frame: Baseline, Week 24 (Epoch 3)
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78
Percent change | -1.24 [-2.50 to -0.45] | -2.04 [-3.36 to -0.88] | -3.52 [-4.62 to -1.87] | -4.37 [-5.36 to -3.37] | -1.67 [-2.61 to -0.27] | -2.51 [-3.94 to -1.32] | -4.06 [-5.52 to -2.87] | -4.47 [-5.49 to -3.48] | -0.63 [-1.56 to 0.37]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p < 0.0001, ANCOVA; Mean Difference (Net) = -1.73, 95% CI 2-sided [-3.17 to -0.29]
Statistical Analysis 2: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p < 0.0001, ANCOVA; Median Difference (Net) = -1.93, 95% CI 2-sided [-3.36 to -0.50]
Statistical Analysis 3: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p < 0.0001, ANCOVA; Mean Difference (Net) = -3.30, 95% CI 2-sided [-4.86 to -1.75]
Statistical Analysis 4: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p < 0.0001, ANCOVA; Mean Difference (Net) = -4.42, 95% CI 2-sided [-5.39 to -3.44]
Statistical Analysis 5: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p < 0.0001, ANCOVA; Mean Difference (Net) = -1.14, 95% CI 2-sided [-2.53 to -0.25]
Statistical Analysis 6: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p < 0.0001, ANCOVA; Mean Difference (Net) = -2.74, 95% CI 2-sided [-4.11 to -1.36]
Statistical Analysis 7: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p < 0.0001, ANCOVA; Mean Difference (Net) = -4.11, 95% CI 2-sided [-5.54 to -2.68]
Statistical Analysis 8: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p < 0.0001, ANCOVA; Mean Difference (Net) = -4.48, 95% CI 2-sided [-5.54 to -3.43]

2. Secondary Outcome: Number of Subjects With Response Rate According to Percent Decrease in Body Weight for Overall Study
Description: Responder rates according to percentage decrease in body weight either ≥ 5 % or ≥ 10 % from baseline
Time Frame: Baseline, Week 24
Population: Full Analysis Set
Measure: Number; unit: Percentage
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 37 | 75 | 78
Percentage
  >=5% | 26.3 | 15.8 | 34.2 | 42.9 | 15.8 | 20.5 | 37.8 | 45.3 | 12.8
  >=10% | 5.3 | 5.3 | 5.3 | 6.5 | 5.3 | 2.6 | 10.8 | 9.3 | 3.8
Statistical Analysis 1: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); >=5%; Test type: Other — Dose finding study; p = 0.099, ANCOVA; Odds Ratio (OR) = 2.38, 95% CI 2-sided [0.85 to 6.67]
Statistical Analysis 2: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); >=5%; Test type: Other — Dose finding study; p = 0.779, ANCOVA; Odds Ratio, log = 1.18, 95% CI 2-sided [0.36 to 3.84]
Statistical Analysis 3: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); >=5%; Test type: Other — Dose finding study; p = 0.011, ANCOVA; Odds Ratio (OR) = 3.69, 95% CI 2-sided [1.35 to 10.11]
Statistical Analysis 4: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); >=5%; Test type: Other — Dose finding study; p < .001, ANCOVA; Odds Ratio (OR) = 5.57, 95% CI 2-sided [2.41 to 12.88]
Statistical Analysis 5: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5%; Test type: Other — Dose finding study; p = 0.812, ANCOVA; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.36 to 3.74]
Statistical Analysis 6: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5%; Test type: Other — Dose finding study; p = 0.229, ANCOVA; Odds Ratio (OR) = 1.94, 95% CI 2-sided [0.66 to 5.69]
Statistical Analysis 7: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5%; Test type: Other — Dose finding study; p = 0.004, ANCOVA; Odds Ratio (OR) = 4.29, 95% CI 2-sided [1.61 to 11.46]
Statistical Analysis 8: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5%; Test type: Other — Dose finding study; p < .001, ANCOVA; Odds Ratio (OR) = 6.37, 95% CI 2-sided [2.72 to 14.93]
Statistical Analysis 9: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); >=10%; Test type: Other — Dose finding study; p = 0.943, ANCOVA; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.10 to 12.41]
Statistical Analysis 10: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); >=10%; Test type: Other — Dose finding study; p = 0.465, ANCOVA; Odds Ratio (OR) = 2.11, 95% CI 2-sided [0.28 to 15.77]
Statistical Analysis 11: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); >=10%; Test type: Other — Dose finding study; p = 0.696, ANCOVA; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.15 to 17.15]
Statistical Analysis 12: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); >=10%; Test type: Other — Dose finding study; p = 0.389, ANCOVA; Odds Ratio (OR) = 2.14, 95% CI 2-sided [0.38 to 12.10]
Statistical Analysis 13: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); >=10%; Test type: Other — Dose finding study; p = 0.976, ANCOVA; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.09 to 11.87]
Statistical Analysis 14: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); >=10%; Test type: Other — Dose finding study; p = 0.986, ANCOVA; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.09 to 11.70]
Statistical Analysis 15: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); >=10%; Test type: Other — Dose finding study; p = 0.181, ANCOVA; Odds Ratio (OR) = 3.51, 95% CI 2-sided [0.56 to 22.18]
Statistical Analysis 16: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); >=10%; Test type: Other — Dose finding study; p = 0.100, ANCOVA; Odds Ratio (OR) = 3.97, 95% CI 2-sided [0.77 to 20.54]

3. Secondary Outcome: Number of Subjects With Response Rate According to Percent Decrease in Body Weight for Subgroups
Description: Responder rates according to percentage decrease in body weight either ≥ 5 % or ≥ 10 % from baseline for dysglycemic, normoglycemic, Type 2 Diabetes Mellitus (T2DM)
Time Frame: Baseline, Week 24
Population: Full Analysis Set
Measure: Number; unit: Percentage
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 37 | 75 | 78
Percentage
  Dysglycemic (>=5%): number analyzed (Participants) | 16 | 16 | 15 | 31 | 15 | 16 | 15 | 31 | 31
  Dysglycemic (>=5%) | 31.3 | 25.0 | 40.0 | 48.4 | 6.7 | 37.5 | 40.0 | 41.9 | 9.7
  Normoglycemic (>=5%): number analyzed (Participants) | 9 | 9 | 9 | 19 | 9 | 9 | 9 | 17 | 20
  Normoglycemic (>=5%) | 44.4 | 11.1 | 44.4 | 47.4 | 11.1 | 11.1 | 55.6 | 52.9 | 20.0
  Type 2 Diabetes Mellitus (T2DM) (>=5%): number analyzed (Participants) | 13 | 13 | 14 | 27 | 14 | 14 | 13 | 27 | 27
  Type 2 Diabetes Mellitus (T2DM) (>=5%) | 7.7 | 15.4 | 28.6 | 37.0 | 28.6 | 14.3 | 30.8 | 44.4 | 14.8
Statistical Analysis 1: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (Dysglycemic); Test type: Other — Dose finding study; p = 0.048, ANCOVA; Odds Ratio (OR) = 6.29, 95% CI 2-sided [1.02 to 38.76]
Statistical Analysis 2: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (Dsyglycemic); Test type: Other — Dose finding study; p = 0.171, ANCOVA; Odds Ratio, log = 3.94, 95% CI 2-sided [0.55 to 28.03]
Statistical Analysis 3: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (Dysglycemic); Test type: Other — Dose finding study; p = 0.041, ANCOVA; Odds Ratio (OR) = 7.17, 95% CI 2-sided [1.09 to 47.27]
Statistical Analysis 4: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (Dysglycemic); Test type: Other — Dose finding study; p = 0.003, ANCOVA; Odds Ratio (OR) = 11.89, 95% CI 2-sided [2.32 to 60.93]
Statistical Analysis 5: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (Dysglycemic); Test type: Other — Dose finding study; p = 0.976, ANCOVA; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.08 to 11.72]
Statistical Analysis 6: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (Dysglycemic); Test type: Other — Dose finding study; p = 0.022, ANCOVA; Odds Ratio (OR) = 8.78, 95% CI 2-sided [1.37 to 56.44]
Statistical Analysis 7: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (Dysglycemic); Test type: Other — Dose finding study; p = 0.032, ANCOVA; Odds Ratio (OR) = 7.50, 95% CI 2-sided [1.20 to 46.99]
Statistical Analysis 8: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (Dysglycemic); Test type: Other — Dose finding study; p = 0.005, ANCOVA; Odds Ratio (OR) = 11.28, 95% CI 2-sided [2.11 to 60.46]
Statistical Analysis 9: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (Normoglycemic); Test type: Other — Dose finding study; p = 0.227, ANCOVA; Odds Ratio (OR) = 3.21, 95% CI 2-sided [0.48 to 21.28]
Statistical Analysis 10: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (Normoglycemic); Test type: Other — Dose finding study; p = 0.763, ANCOVA; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.06 to 7.85]
Statistical Analysis 11: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (Normoglycemic); Test type: Other — Dose finding study; p = 0.095, ANCOVA; Odds Ratio (OR) = 4.68, 95% CI 2-sided [0.76 to 28.70]
Statistical Analysis 12: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (Normoglycemic); Test type: Other — Dose finding study; p = 0.033, ANCOVA; Odds Ratio (OR) = 5.33, 95% CI 2-sided [1.14 to 24.83]
Statistical Analysis 13: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (Normoglycemic); Test type: Other — Dose finding study; p = 0.788, ANCOVA; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.06 to 8.10]
Statistical Analysis 14: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (Normoglycemic); Test type: Other — Dose finding study; p = 0.751, ANCOVA; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.06 to 7.62]
Statistical Analysis 15: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (Normoglycemic); Test type: Other — Dose finding study; p = 0.027, ANCOVA; Odds Ratio (OR) = 8.05, 95% CI 2-sided [1.27 to 51.09]
Statistical Analysis 16: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (Normoglycemic); Test type: Other — Dose finding study; p = 0.023, ANCOVA; Odds Ratio (OR) = 6.64, 95% CI 2-sided [1.30 to 34.00]
Statistical Analysis 17: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (T2DM); Test type: Other — Dose finding study; p = 0.528, ANCOVA; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.05 to 4.78]
Statistical Analysis 18: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (T2DM); Test type: Other — Dose finding study; p = 0.958, ANCOVA; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.17 to 6.68]
Statistical Analysis 19: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (T2DM); Test type: Other — Dose finding study; p = 0.546, ANCOVA; Odds Ratio (OR) = 1.70, 95% CI 2-sided [0.30 to 9.49]
Statistical Analysis 20: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); >=5% (T2DM); Test type: Other — Dose finding test; p = 0.098, ANCOVA; Odds Ratio (OR) = 3.09, 95% CI 2-sided [0.81 to 11.75]
Statistical Analysis 21: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (T2DM); Test type: Other — Dose finding study; p = 0.563, ANCOVA; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.31 to 8.70]
Statistical Analysis 22: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (T2DM); Test type: Other — Dose finding study; p = 0.610, ANCOVA; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.06 to 5.38]
Statistical Analysis 23: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (T2DM); Test type: Other — Dose finding study; p = 0.528, ANCOVA; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.32 to 9.16]
Statistical Analysis 24: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); >=5% (T2DM); Test type: Other — Dose finding study; p = 0.023, ANCOVA; Odds Ratio (OR) = 4.55, 95% CI 2-sided [1.23 to 16.90]

4. Secondary Outcome: Percentage Change From Baseline on Waist Circumference
Description: Waist circumference will be measured to the nearest 0.1cm in a standing position, at the end of a normal expiration, using a tape at the level of the iliac crest.
Time Frame: Baseline, Week 24 (Epoch 3), Week 24 to Week 48 (Epoch 4)
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3) | LIK066 qd/LIK066 25mg qd (Epoch 4) | LIK066 Bid/LIK066 35mg qd (Epoch 4) | Placebo/LIK066 25mg qd (Epoch 4) | Placebo/Placebo (Epoch 4)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78 | 158 | 163 | 39 | 34
Percentage Change | -2.1 [-3.87 to -0.31] | -2.7 [-4.55 to -0.92] | -3.7 [-5.55 to -1.82] | -5.6 [-6.84 to -4.35] | -2.7 [-4.47 to -0.91] | -4.3 [-6.07 to -2.57] | -4.8 [-6.61 to -2.98] | -4.6 [-5.89 to -3.31] | -1.3 [-2.54 to -0.05] | -0.4 [-1.25 to 0.36] | -0.7 [-1.53 to 0.10] | -2.1 [-3.73 to -0.38] | 0.4 [-1.37 to 2.20]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.470, ANCOVA; Median Difference (Net) = -0.8, 95% CI 2-sided [-2.96 to 1.37]
Statistical Analysis 2: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.199, ANCOVA; Median Difference (Net) = -1.4, 95% CI 2-sided [-3.64 to 0.76]
Statistical Analysis 3: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p < 0.001, ANCOVA; Median Difference (Net) = -1.4, 95% CI 2-sided [-3.64 to 0.76]
Statistical Analysis 4: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.206, ANCOVA; Mean Difference (Net) = -1.4, 95% CI 2-sided [-3.56 to 0.77]
Statistical Analysis 5: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.006, ANCOVA; Median Difference (Net) = -3.0, 95% CI 2-sided [-5.18 to -0.88]
Statistical Analysis 6: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.002, ANCOVA; Median Difference (Net) = -3.5, 95% CI 2-sided [-5.70 to -1.30]
Statistical Analysis 7: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p < 0.001, ANCOVA; Mean Difference (Net) = -3.3, 95% CI 2-sided [-5.10 to -1.51]
Statistical Analysis 8: Comparison: LIK066 qd/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Test type: Other — Dose finding study; p = 0.391, ANCOVA; Median Difference (Net) = -0.9, 95% CI 2-sided [-2.82 to 1.10]
Statistical Analysis 9: Comparison: LIK066 Bid/LIK066 35mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Test type: Other — Dose finding study; p = 0.259, ANCOVA; Median Difference (Net) = -2.5, 95% CI 2-sided [-3.10 to 0.84]
Statistical Analysis 10: Comparison: Placebo/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Test type: Other — Dose finding study; p = 0.048, ANCOVA; Mean Difference (Net) = -2.5, 95% CI 2-sided [-4.91 to -0.02]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) in Type 2 Diabetes Mellitus Patients (T2DM)
Description: FPG will be measured from a blood sample obtained after an overnight fast (at least 8h after last evening food intake).
Time Frame: Baseline, Week 24 (Epoch 3), Week 24 to Week 48 (Epoch 4)
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3) | LIK066 qd/LIK066 25mg qd (Epoch 4) | LIK066 Bid/LIK066 35mg qd (Epoch 4) | Placebo/LIK066 25mg qd (Epoch 4) | Placebo/Placebo (Epoch 4)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78 | 158 | 163 | 39 | 34
mmol/L | 1.9 [0.55 to 3.19] | -0.1 [-1.46 to 1.27] | -1.2 [-2.60 to 0.26] | -0.8 [-1.70 to 0.16] | -0.5 [-1.80 to 0.86] | -1.1 [-2.37 to 0.27] | -0.9 [-2.28 to 0.46] | -1.0 [-1.96 to -0.13] | 0.9 [-0.06 to 1.81] | -0.1 [-0.64 to 0.35] | -0.3 [-0.79 to 0.22] | -0.1 [-1.14 to 0.84] | 0.6 [-0.54 to 1.73]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.225, ANCOVA; Mean Difference (Net) = 1.0, 95% CI 2-sided [-0.62 to 2.61]
Statistical Analysis 2: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.247, ANCOVA; Mean Difference (Net) = -1.0, 95% CI 2-sided [-2.62 to 0.68]
Statistical Analysis 3: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.019, ANCOVA; Median Difference (Net) = -2.0, 95% CI 2-sided [-3.75 to -0.34]
Statistical Analysis 4: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.015, ANCOVA; Mean Difference (Net) = -1.6, 95% CI 2-sided [-2.96 to -0.33]
Statistical Analysis 5: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.106, ANCOVA; Mean Difference (Net) = -1.3, 95% CI 2-sided [-2.97 to 0.29]
Statistical Analysis 6: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.020, ANCOVA; Mean Difference (Net) = -1.9, 95% CI 2-sided [-3.54 to -0.31]
Statistical Analysis 7: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.035, ANCOVA; Mean Difference (Net) = -1.8, 95% CI 2-sided [-3.44 to -0.12]
Statistical Analysis 8: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.004, ANCOVA; Mean Difference (Net) = -1.9, 95% CI 2-sided [-3.22 to -0.61]

6. Secondary Outcome: Change From Baseline in Glycated Hemoglobin A1c (HbA1c) in Type 2 Diabetes Mellitus Patients (T2DM)
Description: HbA1c will be measured from a blood sample obtained at indicated visits and will be analyzed at a central laboratory.
Time Frame: Baseline, Week 24 (Epoch 3), Week 24 to week 48 (Epoch 4)
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3) | LIK066 qd/LIK066 25mg qd (Epoch 4) | LIK066 Bid/LIK066 35mg qd (Epoch 4) | Placebo/LIK066 25mg qd (Epoch 4) | Placebo/Placebo (Epoch 4)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78 | 158 | 163 | 39 | 34
mmol/L | 0.1 [-0.23 to 0.45] | -0.5 [-0.82 to -0.13] | -0.9 [-1.24 to -0.50] | -0.7 [-0.92 to -0.44] | -0.3 [-0.68 to 0.00] | -0.5 [-0.83 to -0.15] | -0.6 [-0.98 to -0.28] | -0.6 [-0.87 to -0.40] | -0.3 [-0.50 to -0.02] | 0.2 [0.03 to 0.38] | 0.0 [-0.13 to 0.22] | -0.1 [-0.49 to 0.24] | 0.3 [-0.07 to 0.71]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.082, ANCOVA; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.05 to 0.79]
Statistical Analysis 2: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.319, ANCOVA; Median Difference (Net) = -0.2, 95% CI 2-sided [-0.63 to 0.21]
Statistical Analysis 3: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.008, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.05 to -0.16]
Statistical Analysis 4: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.015, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.76 to -0.08]
Statistical Analysis 5: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.707, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.50 to 0.34]
Statistical Analysis 6: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.280, ANCOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.65 to 0.19]
Statistical Analysis 7: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.086, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.80 to 0.05]
Statistical Analysis 8: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.030, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.72 to -0.04]

7. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) and Mean Sitting Diastolic Blood Pressure (msDBP)
Description: At each study visit (baseline, week 24, Week 48), after the subject has been sitting for 5 minutes with the back supported and both feet placed on the floor, SBP and DBP will be measured
Time Frame: Baseline, Week 24 (Epoch 3) Week 24 to Week 48 (Epoch 4)
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3) | LIK066 qd/LIK066 25mg qd (Epoch 4) | LIK066 Bid/LIK066 35mg qd (Epoch 4) | Placebo/LIK066 25mg qd (Epoch 4) | Placebo/Placebo (Epoch 4)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78 | 158 | 163 | 39 | 34
mmHg
  systolic blood pressure (SBP): number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 37 | 75 | 78 | 58 | 162 | 37 | 34
  systolic blood pressure (SBP) | -1.2 [-4.38 to 1.93] | -1.5 [-4.38 to 1.93] | -4.9 [-8.30 to -1.52] | -1.2 [-3.38 to 1.06] | -0.7 [-3.86 to 2.43] | 0.8 [-2.38 to 3.88] | -2.6 [-5.82 to 0.69] | -1.8 [-4.15 to 0.48] | 1.6 [-0.67 to 3.80] | -0.9 [-2.66 to 0.79] | -1.6 [-3.39 to 0.10] | -5.6 [-9.22 to -2.06] | 0.8 [-2.97 to 4.65]
  diastolic blood pressure (DBP): number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 37 | 75 | 78 | 158 | 162 | 37 | 34
  diastolic blood pressure (DBP) | -0.2 [-2.37 to 2.00] | 0.1 [-2.21 to 2.40] | -2.3 [-4.62 to 0.07] | -1.3 [-2.82 to 0.26] | 0.8 [-1.35 to 3.02] | -1.4 [-3.57 to 0.78] | 0.3 [-1.99 to 2.54] | -1.7 [-3.26 to -0.06] | 0.5 [-1.03 to 2.08] | -0.6 [-1.69 to 0.56] | -1.2 [-2.30 to -0.04] | -2.0 [-4.33 to 0.34] | 0.6 [-1.89 to 3.06]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); SBP; Test type: Other — Dose finding study; p = 0.156, ANCOVA; Mean Difference (Net) = -2.8, 95% CI 2-sided [-6.64 to 1.07]
Statistical Analysis 2: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); SBP; Test type: Other — Dose finding study; p = 0.127, ANCOVA; Mean Difference (Net) = -3.1, 95% CI 2-sided [-7.11 to 0.89]
Statistical Analysis 3: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); SBP; Test type: Other — Dose finding study; p = 0.002, ANCOVA; Mean Difference (Net) = -6.5, 95% CI 2-sided [-10.52 to -2.42]
Statistical Analysis 4: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); SBP; Test type: Other — Dose finding study; p = 0.089, ANCOVA; Mean Difference (Net) = -2.7, 95% CI 2-sided [-5.86 to 0.42]
Statistical Analysis 5: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); SBP; Test type: Other — Dose finding study; p = 0.245, ANCOVA; Mean Difference (Net) = -2.3, 95% CI 2-sided [-6.12 to 1.57]
Statistical Analysis 6: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); SBP; Test type: Other — Dose finding study; p = 0.678, ANCOVA; Mean Difference (Net) = -0.8, 95% CI 2-sided [-4.65 to 3.02]
Statistical Analysis 7: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); SBP; Test type: Other — Dose finding study; p = 0.040, ANCOVA; Mean Difference (Net) = -4.1, 95% CI 2-sided [-8.07 to -0.19]
Statistical Analysis 8: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); SBP; Test type: Other — Dose finding study; p = 0.038, ANCOVA; Mean Difference (Net) = -3.4, 95% CI 2-sided [-6.61 to -0.19]
Statistical Analysis 9: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); DBP; Test type: Other — Dose finding study; p = 0.601, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-3.38 to 1.96]
Statistical Analysis 10: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); DBP; Test type: Other — Dose finding study; p = 0.760, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-3.20 to 2.34]
Statistical Analysis 11: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); DBP; Test type: Other — Dose finding study; p = 0.051, ANCOVA; Mean Difference (Net) = -2.8, 95% CI 2-sided [-5.60 to 0.01]
Statistical Analysis 12: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); DBP; Test type: Other — Dose finding study; p = 0.105, ANCOVA; Mean Difference (Net) = -1.8, 95% CI 2-sided [-3.98 to 0.38]
Statistical Analysis 13: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); DBP; Test type: Other — Dose finding study; p = 0.820, ANCOVA; Mean Difference (Net) = 0.3, 95% CI 2-sided [-2.36 to 2.98]
Statistical Analysis 14: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); DBP; Test type: Other — Dose finding study; p = 0.157, ANCOVA; Mean Difference (Net) = -1.9, 95% CI 2-sided [-4.58 to 0.74]
Statistical Analysis 15: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); DBP; Test type: Other — Dose finding study; p = 0.859, ANCOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-2.99 to 2.49]
Statistical Analysis 16: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); DBP; Test type: Other — Dose finding study; p = 0.054, ANCOVA; Mean Difference (Net) = -2.2, 95% CI 2-sided [-4.41 to 0.04]

8. Secondary Outcome: Change From Baseline in 24-hour Urinary Glucose Excretion
Description: Urinary glucose excretion will be measured from 24-hour urinary collection at indicated visits and will be analyzed at a central laboratory.
Time Frame: Baseline, week 24 (Epoch 3), Week 24 to Week 48 (Epoch 4)
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: mmol/24hr
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3) | LIK066 qd/LIK066 25mg qd (Epoch 4) | LIK066 Bid/LIK066 35mg qd (Epoch 4) | Placebo/LIK066 25mg qd (Epoch 4) | Placebo/Placebo (Epoch 4)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78 | 158 | 163 | 39 | 34
mmol/24hr | 208.6 [101.85 to 315.40] | 134.6 [-8.69 to 277.85] | 377.0 [206.19 to 547.90] | 306.1 [199.59 to 412.62] | 183.0 [32.37 to 333.70] | 193.8 [82.22 to 305.31] | 241.3 [135.13 to 347.30] | 308.9 [198.27 to 419.53] | -17.8 [-94.20 to 58.61] | 26.8 [-30.03 to 83.70] | 122.5 [69.82 to 175.26] | 248.0 [137.72 to 358.33] | -148.9 [-269.62 to -28.10]

9. Secondary Outcome: Percentage Change in Weight in the Overall Population and by Subgroups (Epoch 4)
Description: Between -treatment analysis of percentage change from Week 24 in body weight (kg) at Week 48 (Epoch 4)
Time Frame: Between Week 24 and Week 48 (Epoch 4)
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | LIK066 qd/LIK066 25mg qd (Epoch 4) | LIK066 Bid/LIK066 35mg qd (Epoch 4) | Placebo/LIK066 25mg qd (Epoch 4) | Placebo/Placebo (Epoch 4)
Number analyzed (Participants) | 158 | 163 | 39 | 34
Percentage | -0.2 [-0.70 to 0.33] | -0.2 [-0.68 to 0.35] | -2.4 [-3.47 to -1.33] | 0.4 [-0.74 to 1.55]
Statistical Analysis 1: Comparison: LIK066 qd/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Test type: Other — Dose finding study; p = 0.355, ANCOVA; Median Difference (Net) = -0.6, 95% CI 2-sided [-1.84 to 0.66]
Statistical Analysis 2: Comparison: LIK066 Bid/LIK066 35mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Test type: Other — Dose finding study; p = 0.373, ANCOVA; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.83 to 0.69]
Statistical Analysis 3: Comparison: Placebo/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Test type: Other — Dose finding study; p < 0.001, ANCOVA; Mean Difference (Net) = -2.8, 95% CI 2-sided [-4.36 to -1.24]

10. Secondary Outcome: Change From Baseline to Week 24 (Epoch 3) in the 24-hour Urinary Calcium Excretion
Description: Evaluation of 24-hour urinary calcium excretion after 24 week of treatment.
Time Frame: Baseline, Week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmol/24hr
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78
mmol/24hr
  Baseline: number analyzed (Participants) | 12 | 9 | 9 | 16 | 9 | 13 | 38 | 20 | 26
  Baseline | 49.6 (25.08) | 33.1 (29.65) | 40.2 (21.55) | 34.6 (17.56) | 44.7 (26.83) | 43.6 (16.91) | 38.0 (22.13) | 47.9 (23.64) | 43.0 (22.63)
  Week 24 (Timepoint 1): number analyzed (Participants) | 38 | 38 | 38 | 77 | 5 | 12 | 8 | 15 | 23
  Week 24 (Timepoint 1) | 48.8 (26.59) | 38.1 (32.20) | 39.8 (22.48) | 40.1 (18.20) | 52.4 (32.78) | 45.9 (15.41) | 38.0 (22.13) | 48.1 (21.93) | 44.7 (23.0)
  Week 24 (Timepoint 2): number analyzed (Participants) | 10 | 7 | 7 | 8 | 5 | 12 | 8 | 15 | 23
  Week 24 (Timepoint 2) | 54.2 (29.34) | 42.0 (29.99) | 39.2 (20.24) | 62.8 (34.26) | 51.2 (35.32) | 54.6 (23.77) | 37.9 (32.33) | 53.0 (26.95) | 52.2 (30.75)
  Week 24 (Timepoint 3): number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 15 | 23
  Week 24 (Timepoint 3) | 5.4 (22.74) | 3.9 (19.56) | -0.6 (12.07) | 22.8 (28.42) | -1.2 (7.77) | 8.7 (18.21) | -0.1 (14.39) | 4.9 (26.20) | 7.5 (32.91)

11. Secondary Outcome: Change From Baseline Week 24 to Week 48 (Epoch 4) in the 24-hour Urinary Calcium Excretion
Description: Evaluation of 24-hour urinary calcium after 48 weeks of treatment
Time Frame: Baseline, Week 24, Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmol/24hr
Arm/Group | LIK066 qd/LIK066 25mg qd (Epoch 4) | LIK066 Bid/LIK066 35mg qd (Epoch 4) | Placebo/LIK066 25mg qd (Epoch 4) | Placebo/Placebo (Epoch 4)
Number analyzed (Participants) | 158 | 163 | 39 | 34
mmol/24hr
  Baseline: number analyzed (Participants) | 33 | 40 | 11 | 13
  Baseline | 4.8 (3.02) | 5.0 (2.84) | 4.6 (0.91) | 5.6 (4.07)
  Week 48(Timepoint 1): number analyzed (Participants) | 26 | 33 | 10 | 9
  Week 48(Timepoint 1) | 5.1 (307) | 5.2 (2.95) | 4.5 (0.95) | 6.6 (4.55)
  Week 48(Timepoint 2): number analyzed (Participants) | 26 | 33 | 10 | 9
  Week 48(Timepoint 2) | 4.6 (2.33) | 5.6 (4.55) | 5.4 (3.65) | 4.8 (2.10)
  Week 48(Timepoint 3): number analyzed (Participants) | 26 | 33 | 10 | 9
  Week 48(Timepoint 3) | -0.5 (3.41) | 0.4 (2.81) | 0.9 (4.10) | -1.8 (3.26)

12. Secondary Outcome: Change From Baseline to Week 24 (Epoch 3) in the 24-hour Urinary Phosphorus Excretion
Description: Evaluation of 24-hour urinary phosphorus excretion after 24 weeks of treatment
Time Frame: Week 24, Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmol/24hr
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78
mmol/24hr
  Baseline: number analyzed (Participants) | 12 | 10 | 10 | 16 | 9 | 14 | 9 | 21 | 26
  Baseline | 282.1 (128.10) | 240.5 (74.64) | 254.5 (105.70) | 291.5 (175.10) | 284.0 (117.60) | 241.8 (82.75) | 277.0 (99.67) | 293.7 (120.70) | 297.0 (145.10)
  Week 24 (Timepoint 1): number analyzed (Participants) | 10 | 7 | 8 | 10 | 6 | 13 | 8 | 16 | 24
  Week 24 (Timepoint 1) | 284.0 (140.10) | 239.7 (80.40) | 260.9 (111.10) | 275.0 (101.30) | 319.9 (32.78) | 246.5 (84.19) | 299.3 (79.06) | 302.5 (121.30) | 307.9 (145.90)
  Week 24 (Timepoint 2): number analyzed (Participants) | 10 | 7 | 8 | 10 | 6 | 13 | 8 | 16 | 24
  Week 24 (Timepoint 2) | 297.7 (117.40) | 295.3 (95.60) | 299.2 (145.50) | 264.7 (74.84) | 317.8 (205.10) | 341.6 (109.20) | 260.5 (124.80) | 289.3 (83.62) | 352.8 (159.30)
  Week 24 (Timepoint 3): number analyzed (Participants) | 10 | 7 | 8 | 10 | 6 | 13 | 8 | 16 | 24
  Week 24 (Timepoint 3) | 13.0 (132.00) | 55.6 (89.81) | 38.3 (70.00) | -10.2 (103.60) | -2.1 (159.60) | 95.1 (67.36) | -38.7 (107.80) | -13.2 (153.80) | 44.9 (177.60)

13. Secondary Outcome: Change From Baseline Week 24 to Week 48 (Epoch 4) in the 24-hour Urinary Phosphorus Excretion
Description: Evaluation of 24-hour urinary phosphorus excretion after 48 weeks of treatment
Time Frame: Week 24, Week 48
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mmol/24hr
Arm/Group | LIK066 qd/LIK066 25mg qd (Epoch 4) | LIK066 Bid/LIK066 35mg qd (Epoch 4) | Placebo/LIK066 25mg qd (Epoch 4) | Placebo/Placebo (Epoch 4)
Number analyzed (Participants) | 158 | 163 | 39 | 34
mmol/24hr
  Baseline: number analyzed (Participants) | 36 | 42 | 12 | 13
  Baseline | 27.6 (11.46) | 30.5 (11.63) | 28.6 (14.11) | 40.2 (15.96)
  Week 48 (Timepoint 1): number analyzed (Participants) | 30 | 35 | 12 | 9
  Week 48 (Timepoint 1) | 27.5 (11.73) | 30.2 (11.85) | 28.6 (14.11) | 44.4 (17.60)
  Week 48 (Timepoint 2): number analyzed (Participants) | 30 | 35 | 12 | 9
  Week 48 (Timepoint 2) | 24.7 (12.74) | 31.1 (16.21) | 31.0 (14.67) | 29.0 (15.42)
  Week 48(Timepoint 3): number analyzed (Participants) | 30 | 35 | 12 | 9
  Week 48(Timepoint 3) | -2.8 (11.44) | 0.9 (14.52) | 2.4 (17.33) | -15.5 (18.92)

14. Secondary Outcome: Change From Baseline in Fasting Lipid Profile (Lipoproteins)
Description: Between-treatment analysis of change after 24 weeks of treatment and between Week 24 and Week 48
Time Frame: Baseline, Week 24, Week 24 to Week 48 (Epoch 4)
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: g/L
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3) | LIK066 qd/LIK066 25mg qd (Epoch 4) | LIK066 Bid/LIK066 35mg qd (Epoch 4) | Placebo/LIK066 25mg qd (Epoch 4) | Placebo/Placebo (Epoch 4)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78 | 158 | 163 | 39 | 34
g/L
  Apoliprotein A1: number analyzed (Participants) | 37 | 38 | 32 | 77 | 36 | 38 | 35 | 71 | 78 | 151 | 152 | 36 | 34
  Apoliprotein A1 | 8.9 [4.26 to 13.61] | 8.13 [3.27 to 13.30] | 10.7 [5.38 to 15.97] | 8.9 [5.55 to 12.21] | 5.3 [0.487 to 10.17] | 8.1 [3.44 to 12.86] | 6.7 [1.75 to 11.59] | 11.0 [7.47 to 14.44] | 6.7 [3.41 to 10.06] | 3.0 [0.92 to 5.10] | 3.4 [1.22 to 5.51] | 5.6 [1.35 to 9.89] | -0.7 [-5.27 to 3.87]
  Apoliprotein B: number analyzed (Participants) | 37 | 38 | 32 | 77 | 36 | 38 | 35 | 75 | 78 | 151 | 152 | 36 | 34
  Apoliprotein B | 2.9 [-5.32 to 11.08] | 7.7 [-1.23 to 16.61] | 3.3 [-6.06 to 12.72] | 12.4 [6.57 to 18.32] | -0.4 [-8.91 to 8.18] | 4.5 [-3.84 to 12.74] | 2.3 [-6.36 to 10.98] | 3.9 [-2.29 to 10.01] | 5.8 [-0.03 to 11.69] | -1.7 [-4.39 to 1.08] | -2.4 [-5.23 to 0.38] | -2.3 [-7.85 to 3.31] | -2.0 [-8.00 to 3.96]

15. Secondary Outcome: Change From Baseline in High Sensitive C-reactive Protein (hsCRP)
Description: Between-treatment analysis of change after 24 weeks of treatment and between Week 24 and Week 48
Time Frame: Baseline to Week 24, Week 24 to Week 48 (Epoch 4)
Population: Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3) | LIK066 qd/LIK066 25mg qd (Epoch 4) | LIK066 Bid/LIK066 35mg qd (Epoch 4) | Placebo/LIK066 25mg qd (Epoch 4) | Placebo/Placebo (Epoch 4)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78 | 158 | 163 | 39 | 34
mg/L | 0.99 [0.78 to 1.25] | 1.06 [0.83 to 1.36] | 1.31 [1.01 to 1.69] | 0.98 [0.83 to 1.16] | 1.02 [0.80 to 1.30] | 0.93 [0.74 to 118] | 1.00 [0.78 to 1.27] | 0.98 [0.83 to 1.17] | 0.92 [0.78 to 1.09] | 0.95 [0.85 to 1.06] | 0.93 [0.83 to 1.04] | 0.96 [0.77 to 1.20] | 1.07 [0.84 to 1.36]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.632, ANCOVA; Mean Difference (Net) = 1.07, 95% CI 2-sided [0.81 to 1.42]
Statistical Analysis 2: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.352, ANCOVA; Mean Difference (Net) = 1.15, 95% CI 2-sided [0.86 to 1.55]
Statistical Analysis 3: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.027, ANCOVA; Mean Difference (Net) = 1.41, 95% CI 2-sided [1.04 to 1.92]
Statistical Analysis 4: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.587, ANCOVA; Mean Difference (Net) = 1.07, 95% CI 2-sided [0.85 to 1.35]
Statistical Analysis 5: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.508, ANCOVA; Mean Difference (Net) = 1.10, 95% CI 2-sided [0.82 to 1.47]
Statistical Analysis 6: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.945, ANCOVA; Mean Difference (Net) = 1.01, 95% CI 2-sided [0.76 to 1.34]
Statistical Analysis 7: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); Test type: Other — Dose finding study; p = 0.602, ANCOVA; Mean Difference (Net) = 1.08, 95% CI 2-sided [0.81 to 1.45]
Statistical Analysis 8: Comparison: LIK066 50mg Bid (Epoch 3); Test type: Other — Dose finding study; p = 0.612, ANCOVA; Mean Difference (Net) = 1.06, 95% CI 2-sided [0.84 to 1.35]
Statistical Analysis 9: Comparison: LIK066 qd/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Test type: Other — Dose finding study; p = 0.382, ANCOVA; Median Difference (Net) = 0.89, 95% CI 2-sided [0.68 to 1.16]
Statistical Analysis 10: Comparison: LIK066 Bid/LIK066 35mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Test type: Other — Dose finding study; p = 0.310, ANCOVA; Median Difference (Net) = 0.87, 95% CI 2-sided [0.67 to 1.14]
Statistical Analysis 11: Comparison: Placebo/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Test type: Other — Dose finding study; p = 0.525, ANCOVA; Mean Difference (Net) = 0.90, 95% CI 2-sided [0.65 to 1.25]

16. Secondary Outcome: Change From Baseline in Fasting Lipid Profile (Triglycerides/Cholesterol)
Description: Between-treatment analysis of change after 24 weeks of treatment and between Week 24 and Week 48
Time Frame: Baseline to Week 24, Week 24 to Week 48 (Epoch 4)
Population: Full Analysis Set
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3) | Placebo (Epoch 3) | LIK066 qd/LIK066 25mg qd (Epoch 4) | LIK066 Bid/LIK066 35mg qd (Epoch 4) | Placebo/LIK066 25mg qd (Epoch 4) | Placebo/Placebo (Epoch 4)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 38 | 76 | 78 | 158 | 163 | 39 | 34
mmol/L
  Triglycerides (TG): number analyzed (Participants) | 37 | 38 | 32 | 77 | 37 | 38 | 38 | 71 | 78 | 150 | 149 | 36 | 34
  Triglycerides (TG) | -3.8 [-14.91 to 7.26] | 1.3 [-11.19 to 13.80] | -11.5 [-24.03 to .093] | -3.0 [-10.94 to 4.91] | 2.3 [-8.94 to 13.57] | 1.7 [-9.30 to 12.77] | 5.5 [-5.94 to 16.89] | -7.4 [-15.60 to 0.87] | 4.0 [-3.82 to 11.87] | 6.7 [0.18 to 13.13] | 12.4 [5.75 to 19.13] | -0.9 [-14.48 to 12.59] | 4.8 [-9.57 to 19.16]
  Total Cholesterol (TC): number analyzed (Participants) | 37 | 38 | 32 | 77 | 36 | 38 | 35 | 71 | 78 | 151 | 152 | 36 | 34
  Total Cholesterol (TC) | 6.0 [-0.92 to 12.99] | 7.3 [-0.23 to 14.92] | 4.8 [-3.15 to 12.78] | 14.6 [9.61 to 19.58] | 1.5 [-5.79 to 8.71] | 5.1 [-1.89 to 12.19] | 6.4 [-0.94 to 13.75] | 8.8 [-0.23 to 9.70] | 4.7 [-0.23 to 9.70] | 0.8 [-1.65 to 3.27] | 0.3 [-2.22 to 2.81] | 0.8 [-4.22 to 5.81] | -1.7 [-7.04 to 3.68]
  HDL Cholesterol: number analyzed (Participants) | 37 | 38 | 32 | 77 | 36 | 38 | 35 | 71 | 78 | 151 | 152 | 36 | 34
  HDL Cholesterol | 0.8 [-5.25 to 6.76] | 4.9 [-1.52 to 11.28] | 5.2 [-1.55 to 12.01] | 8.0 [3.71 to 12.25] | 2.9 [-3.29 to 9.16] | 2.4 [-3.60 to 8.48] | 1.5 [-4.86 to 7.81] | 8.0 [3.56 to 12.47] | 0.7 [-3.54 to 5.00] | 3.9 [0.84 to 7.03] | 3.7 [0.54 to 6.90] | 9.2 [2.88 to 15.57] | 0.7 [-6.11 to 7.48]
  LDL Cholesterol: number analyzed (Participants) | 37 | 38 | 32 | 77 | 36 | 38 | 35 | 71 | 78 | 151 | 152 | 36 | 34
  LDL Cholesterol | 8.7 [-2.14 to 19.61] | 17.5 [5.73 to 29.20] | 8.2 [-4.21 to 20.25] | 21.8 [14.08 to 29.55] | 4.1 [-7.22 to 15.38] | 8.7 [-2.26 to 19.68] | 7.7 [-3.77 to 19.13] | 10.9 [2.80 to 19.04] | 12.5 [4.70 to 20.30] | -0.6 [-4.14 to 2.96] | -1.2 [-4.79 to 2.49] | -1.4 [-8.66 to 5.83] | -3.5 [-11.28 to 4.24]
Statistical Analysis 1: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); Triglycerides (TG); Test type: Other — Dose finding study; p = 0.254, ANCOVA; Mean Difference (Net) = -7.9, 95% CI 2-sided [-21.37 to 5.65]
Statistical Analysis 2: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); Triglycerides (TG); Test type: Other — Dose finding study; p = 0.716, ANCOVA; Mean Difference (Net) = -2.7, 95% CI 2-sided [-17.44 to 11.99]
Statistical Analysis 3: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); Triglycerides (TG); Test type: Other — Dose finding study; p = 0.038, ANCOVA; Mean Difference (Net) = -15.6, 95% CI 2-sided [-30.30 to -0.86]
Statistical Analysis 4: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); Triglycerides (TG); Test type: Other — Dose finding study; p = 0.213, ANCOVA; Mean Difference (Net) = -7.0, 95% CI 2-sided [-18.15 to 4.06]
Statistical Analysis 5: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); Triglycerides (TG); Test type: Other — Dose finding study; p = 0.806, ANCOVA; Mean Difference (Net) = -1.7, 95% CI 2-sided [-15.38 to 11.96]
Statistical Analysis 6: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); Triglycerides (TG); Test type: Other — Dose finding study; p = 0.739, ANCOVA; Mean Difference (Net) = -2.3, 95% CI 2-sided [-15.80 to 11.21]
Statistical Analysis 7: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); Triglycerides (TG); Test type: Other — Dose finding study; p = 0.837, ANCOVA; Mean Difference (Net) = 1.4, 95% CI 2-sided [-12.36 to 15.26]
Statistical Analysis 8: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); Triglycerides (TG); Test type: Other; p = 0.049, ANCOVA; Mean Difference (Net) = -11.4, 95% CI 2-sided [-22.71 to -0.07]
Statistical Analysis 9: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); Total Cholesterol (TC); Test type: Other — Dose finding study; p = 0.764, ANCOVA; Median Difference (Net) = 1.3, 95% CI 2-sided [-7.22 to 9.82]
Statistical Analysis 10: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); Total Cholesterol (TC); Test type: Other — Dose finding study; p = 0.571, ANCOVA; Mean Difference (Net) = 2.6, 95% CI 2-sided [-6.43 to 11.63]
Statistical Analysis 11: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); Total Cholesterol (TC); Test type: Other — Dose finding study; p = 0.987, ANCOVA; Mean Difference (Net) = 0.1, 95% CI 2-sided [-9.30 to 9.46]
Statistical Analysis 12: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); Total Cholesterol (TC); Test type: Other — Dose finding study; p = 0.006, ANCOVA; Mean Difference (Net) = 9.9, 95% CI 2-sided [2.85 to 16.87]
Statistical Analysis 13: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); Total Cholesterol (TC); Test type: Other — Dose finding study; p = 0.463, ANCOVA; Mean Difference (Net) = -3.3, 95% CI 2-sided [-12.03 to 5.48]
Statistical Analysis 14: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); Total Cholesterol (TC); Test type: Other — Dose finding study; p = 0.925, ANOVA; Mean Difference (Net) = 0.4, 95% CI 2-sided [-8.18 to 9.01]
Statistical Analysis 15: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); Total Cholesterol (TC); Test type: Other — Dose finding study; p = 0.711, ANCOVA; Mean Difference (Net) = 1.7, 95% CI 2-sided [-7.19 to 10.53]
Statistical Analysis 16: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); Total Cholesterol (TC); Test type: Other — Dose finding study; p = 0.265, ANCOVA; Mean Difference (Net) = 4.1, 95% CI 2-sided [-3.10 to 11.26]
Statistical Analysis 17: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); HDL Cholesterol; Test type: Other — Dose finding study; p = 0.995, ANCOVA; Median Difference (Net) = 0.0, 95% CI 2-sided [-7.31 to 7.36]
Statistical Analysis 18: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); HDL Cholesterol; Test type: Other — Dose finding study; p = 0.288, ANCOVA; Mean Difference (Net) = 4.1, 95% CI 2-sided [-3.52 to 11.81]
Statistical Analysis 19: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); HDL Cholesterol; Test type: Other — Dose finding study; p = 0.269, ANCOVA; Mean Difference (Net) = 4.5, 95% CI 2-sided [-3.50 to 12.50]
Statistical Analysis 20: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); HDL Cholesterol; Test type: Other — Dose finding study; p = 0.018, ANCOVA; Median Difference (Net) = 7.3, 95% CI 2-sided [1.23 to 13.27]
Statistical Analysis 21: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); HDL Cholesterol; Test type: Other — Dose finding study; p = 0.565, ANCOVA; Median Difference (Net) = 2.2, 95% CI 2-sided [-5.32 to 9.73]
Statistical Analysis 22: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); HDL Cholesterol; Test type: Other — Dose finding study; p = 0.649, ANCOVA; Mean Difference (Net) = 1.7, 95% CI 2-sided [-5.67 to 9.09]
Statistical Analysis 23: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); HDL Cholesterol; Test type: Other — Dose finding study; p = 0.847, ANCOVA; Mean Difference (Net) = 0.7, 95% CI 2-sided [-6.87 to 8.36]
Statistical Analysis 24: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); HDL Cholesterol; Test type: Other — Dose finding study; p = 0.020, ANCOVA; Mean Difference (Net) = 7.3, 95% CI 2-sided [1.14 to 13.43]
Statistical Analysis 25: Comparison: LIK066 2.5mg qd (Epoch 3) vs Placebo (Epoch 3); LDL Cholesterol; Test type: Other — Dose finding study; p = 0.579, ANCOVA; Mean Difference (Net) = -3.8, 95% CI 2-sided [-17.09 to 9.57]
Statistical Analysis 26: Comparison: LIK066 10mg qd (Epoch 3) vs Placebo (Epoch 3); LDL Cholesterol; Test type: Other; p = 0.487, ANCOVA; Mean Difference (Net) = 5.0, 95% CI 2-sided [-9.08 to 19.02]
Statistical Analysis 27: Comparison: LIK066 50mg qd (Epoch 3) vs Placebo (Epoch 3); LDL Cholesterol; Test type: Other — Dose finding study; p = 0.561, ANCOVA; Mean Difference (Net) = -4.3, 95% CI 2-sided [-18.96 to 10.30]
Statistical Analysis 28: Comparison: LIK066 150mg qd (Epoch 3) vs Placebo (Epoch 3); LDL Cholesterol; Test type: Other; p = 0.097, ANCOVA; Mean Difference (Net) = 9.3, 95% CI 2-sided [-1.68 to 20.25]
Statistical Analysis 29: Comparison: LIK066 2.5mg Bid (Epoch 3) vs Placebo (Epoch 3); LDL Cholesterol; Test type: Other — Dose finding study; p = 0.227, ANCOVA; Mean Difference (Net) = -8.4, 95% CI 2-sided [-22.10 to 5.26]
Statistical Analysis 30: Comparison: LIK066 5mg Bid (Epoch 3) vs Placebo (Epoch 3); LDL Cholesterol; Test type: Other — Dose finding study; p = 0.580, ANCOVA; Mean Difference (Net) = -3.8, 95% CI 2-sided [-17.22 to 9.64]
Statistical Analysis 31: Comparison: LIK066 25mg Bid (Epoch 3) vs Placebo (Epoch 3); LDL Cholesterol; Test type: Other — Dose finding study; p = 0.494, ANCOVA; Mean Difference (Net) = -4.8, 95% CI 2-sided [-18.67 to 9.03]
Statistical Analysis 32: Comparison: LIK066 50mg Bid (Epoch 3) vs Placebo (Epoch 3); LDL Cholesterol; Test type: Other — Dose finding study; p = 0.782, ANCOVA; Mean Difference (Net) = -1.6, 95% CI 2-sided [-12.81 to 9.65]
Statistical Analysis 33: Comparison: LIK066 qd/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Triglycerides (TG); Test type: Other — Dose finding study; p = 0.816, ANCOVA; Mean Difference (Net) = 1.9, 95% CI 2-sided [-13.82 to 17.54]
Statistical Analysis 34: Comparison: LIK066 Bid/LIK066 35mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Triglycerides (TG); Test type: Other — Dose finding study; p = 0.341, ANCOVA; Mean Difference (Net) = 8.02, 95% CI 2-sided [-8.13 to 23.42]
Statistical Analysis 35: Comparison: Placebo/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Triglycerides (TG); Test type: Other — Dose finding study; p = 0.566, ANCOVA; Median Difference (Net) = 9.99, 95% CI 2-sided [-25.39 to 13.91]
Statistical Analysis 36: Comparison: LIK066 qd/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Total Cholesterol (TC); Test type: Other — Dose finding study; p = 0.405, ANCOVA; Mean Difference (Net) = 2.98, 95% CI 2-sided [-3.38 to 8.36]
Statistical Analysis 37: Comparison: LIK066 Bid/LIK066 35mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Total Cholesterol (TC); Test type: Other — Dose finding study; p = 0.511, ANCOVA; Median Difference (Net) = 2.0, 95% CI 2-sided [-3.92 to 7.87]
Statistical Analysis 38: Comparison: Placebo/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); Total Cholesterol (TC); Test type: Other — Dose finding study; p = 0.506, ANCOVA; Mean Difference (Net) = 2.5, 95% CI 2-sided [-4.83 to 9.79]
Statistical Analysis 39: Comparison: LIK066 qd/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); HDL Cholesterol; Test type: Other — Dose finding study; p = 0.392, ANCOVA; Median Difference (Net) = 3.3, 95% CI 2-sided [-4.20 to 10.70]
Statistical Analysis 40: Comparison: LIK066 Bid/LIK066 35mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); HDL Cholesterol; Test type: Other — Dose finding study; p = 0.426, ANOVA; Mean Difference (Net) = 3.0, 95% CI 2-sided [-4.45 to 10.53]
Statistical Analysis 41: Comparison: Placebo/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); HDL Cholesterol; Test type: Other — Dose finding study; p = 0.071, ANCOVA; Mean Difference (Net) = 8.5, 95% CI 2-sided [-0.72 to 17.80]
Statistical Analysis 42: Comparison: LIK066 qd/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); LDL Cholesterol; Test type: Other — Dose finding study; p = 0.498, ANCOVA; Mean Difference (Net) = 2.9, 95% CI 2-sided [-5.56 to 11.42]
Statistical Analysis 43: Comparison: LIK066 Bid/LIK066 35mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); LDL Cholesterol; Test type: Other — Dose finding study; p = 0.586, ANCOVA; Median Difference (Net) = 2.4, 95% CI 2-sided [-6.17 to 10.90]
Statistical Analysis 44: Comparison: Placebo/LIK066 25mg qd (Epoch 4) vs Placebo/Placebo (Epoch 4); LDL Cholesterol; Test type: Other — Dose finding study; p = 0.696, ANCOVA; Mean Difference (Net) = 2.1, 95% CI 2-sided [-8.47 to 12.67]

17. Secondary Outcome: Pharmacokinetics of LIK066: Observe Maximum Plasma Concentration (Cmax)
Description: Observe maximum plasma concentration following administration of LIK066 (Cmax)
Time Frame: Summary at Week 24 from qd or bid regimens
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 37 | 76
ng/mL | 80.0 (97.2) | 128 (00.0) | 798 (397) | 1810 (545) | 38.6 (5.22) | 84.2 (19.0) | 523 (118) | 811 (367)

18. Secondary Outcome: Pharmacokinetics of LIK066: Time to Reach the Maximum Concentration (Tmax)
Description: Time to reach the maximum concentration after administration of LIK066 (Tmax)
Time Frame: Summary at Week 24 for qd or bid regimens
Population: Full Analysis Set
Measure: Median (Full Range); unit: hour
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 37 | 76
hour | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 1.00] | 1.01 [1.00 to 2.08] | 1.02 [1.00 to 2.00] | 1.00 [0.983 to 1.00] | 1.00 [0.917 to 2.00] | 0.992 [0.900 to 1.00] | 1.00 [0.983 to 2.00]

19. Secondary Outcome: Pharmacokinetics of LIK066: Area Under the Plasma Concentration-time Curve From Time Zero Time 't' (AUC0-t)
Description: Area under the plasma concentration-time curve from time zero time 't' where t is a defined time point after administration (AUC0-t)
Time Frame: Summary at Week 24 from qd or bid regimens (0-6h)
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 37 | 76
hr*ng/mL | 196 (186) | 275 (000) | 2280 (522) | 5700 (1490) | 105 (17.1) | 273 (69.3) | 1520 (277) | 2190 (841)

20. Secondary Outcome: Pharmacokinetics of LIK066: Last Non-zero Concentration Area Under the Curve (AUClast)
Description: Last non-zero concentration area under the curve (AUClast)
Time Frame: Summary at Week 24 from qd or bid regimens
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | LIK066 2.5mg qd (Epoch 3) | LIK066 10mg qd (Epoch 3) | LIK066 50mg qd (Epoch 3) | LIK066 150mg qd (Epoch 3) | LIK066 2.5mg Bid (Epoch 3) | LIK066 5mg Bid (Epoch 3) | LIK066 25mg Bid (Epoch 3) | LIK066 50mg Bid (Epoch 3)
Number analyzed (Participants) | 38 | 38 | 38 | 77 | 38 | 39 | 37 | 76
hr*ng/mL | 196 (186) | 275 (000) | 2290 (526) | 5690 (1480) | 105 (17.2) | 273 (70.2) | 1520 (271) | 2190 (843)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment, plus 30 days post treatment, up to maximum duration of approximately 15 months.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Groups:
- LIK066 2.5 mg qd (Epoch 3)/25 mg qd (Epoch 4): LIK066 2.5mg qd (once daily) dosing frequency for 24 weeks (Epoch3), then LIK066 25 mg qd for 24 weeks (Epoch 4)
- LIK066 10 mg qd/25 mg qd: LIK066 10mg qd (once daily) dosing frequency for 24 weeks
- LIK066 50 mg qd/25 mg qd: LIK066 50mg qd (once daily) dosing frequency for 24 weeks
- LIK066 150 mg qd/25 mg qd: LIK066 150mg qd (once daily) dosing frequency for 24 weeks
- LIK066 2.5 mg Bid/35 mg qd: LIK066 2.5mg bid (twice daily) dosing frequency for 24 weeks
- LIK066 5 mg Bid/35 mg qd: LIK066 5mg bid (twice daily) dosing frequency for 24 weeks
- LIK066 25 mg Bid/35 mg qd: LIK066 25mg bid (twice daily) dosing frequency for 24 weeks
- LIK066 50 mg Bid/35 mg qd: LIK066 50mg bid (twice daily) dosing frequency for 24 weeks
- Placebo/Placebo: Matching placebo tablets
Arm/Group | LIK066 2.5 mg qd (Epoch 3)/25 mg qd (Epoch 4) | LIK066 10 mg qd/25 mg qd | LIK066 50 mg qd/25 mg qd | LIK066 150 mg qd/25 mg qd | LIK066 2.5 mg Bid/35 mg qd | LIK066 5 mg Bid/35 mg qd | LIK066 25 mg Bid/35 mg qd | LIK066 50 mg Bid/35 mg qd | Placebo/LIK066 25 mg qd (Epoch 4) | Placebo/Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 1/38 | 0/38 | 0/77 | 1/38 | 0/39 | 0/38 | 0/76 | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 3/38 | 3/38 | 1/38 | 3/77 | 5/38 | 2/39 | 2/38 | 1/76 | 1/40 | 4/38
Other Adverse Events (participants affected / at risk) | 33/38 | 24/38 | 24/38 | 55/77 | 31/38 | 32/39 | 26/38 | 47/76 | 32/40 | 32/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LIK066 2.5 mg qd (Epoch 3)/25 mg qd (Epoch 4) (N=38) | LIK066 10 mg qd/25 mg qd (N=38) | LIK066 50 mg qd/25 mg qd (N=38) | LIK066 150 mg qd/25 mg qd (N=77) | LIK066 2.5 mg Bid/35 mg qd (N=38) | LIK066 5 mg Bid/35 mg qd (N=39) | LIK066 25 mg Bid/35 mg qd (N=38) | LIK066 50 mg Bid/35 mg qd (N=76) | Placebo/LIK066 25 mg qd (Epoch 4) (N=40) | Placebo/Placebo (N=38)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Breast enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LIK066 2.5 mg qd (Epoch 3)/25 mg qd (Epoch 4) (N=38) | LIK066 10 mg qd/25 mg qd (N=38) | LIK066 50 mg qd/25 mg qd (N=38) | LIK066 150 mg qd/25 mg qd (N=77) | LIK066 2.5 mg Bid/35 mg qd (N=38) | LIK066 5 mg Bid/35 mg qd (N=39) | LIK066 25 mg Bid/35 mg qd (N=38) | LIK066 50 mg Bid/35 mg qd (N=76) | Placebo/LIK066 25 mg qd (Epoch 4) (N=40) | Placebo/Placebo (N=38)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Microvascular coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Porokeratosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type IIa hyperlipidaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inner ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye movement disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myopic chorioretinal degeneration (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 3 | 7 | 3 | 3 | 0 | 0 | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 4 | 8 | 9 | 5 | 4 | 6 | 6 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2 | 3 | 1 | 3 | 2 | 2 | 1 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 4 | 7 | 7 | 3 | 4 | 4 | 4 | 4
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 6 | 7 | 6 | 11 | 12 | 5 | 8 | 8 | 7 | 9
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 4 | 7 | 5 | 1 | 4 | 3 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 14 | 7 | 15 | 42 | 16 | 12 | 14 | 29 | 14 | 8
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyschezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 10 | 5 | 4 | 6 | 3 | 10
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 1 | 2 | 5 | 5 | 1 | 3 | 4 | 2 | 2
Faeces hard (Gastrointestinal disorders) | 2 | 2 | 2 | 3 | 5 | 0 | 2 | 2 | 1 | 3
Flatulence (Gastrointestinal disorders) | 7 | 9 | 9 | 21 | 12 | 6 | 11 | 21 | 6 | 8
Frequent bowel movements (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 2 | 2 | 4 | 3 | 7 | 0 | 3 | 2 | 0 | 4
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 1 | 4 | 5 | 4 | 1 | 4 | 3 | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 2 | 3 | 1 | 4 | 1 | 3
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 3 | 8 | 3 | 3 | 4 | 5 | 5
Splenic artery aneurysm (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hunger (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Thirst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial vulvovaginitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balanitis candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 4 | 0 | 2 | 2 | 0 | 2 | 2 | 2 | 3 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genital candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 3 | 5 | 2 | 2 | 3 | 1 | 2
Nasopharyngitis (Infections and infestations) | 4 | 2 | 3 | 8 | 4 | 3 | 7 | 5 | 0 | 2
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis externa fungal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0
Sinobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 3 | 1 | 1 | 0 | 1 | 3 | 3 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 3 | 7 | 2 | 2 | 1 | 2 | 5 | 5
Urinary tract infection (Infections and infestations) | 3 | 1 | 3 | 1 | 1 | 4 | 4 | 4 | 2 | 5
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 3
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 4 | 2 | 0 | 1 | 1 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Apolipoprotein A-I decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood albumin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 0
Blood glucose increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine urine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram change (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glomerular filtration rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin urine present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
High density lipoprotein decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Liver scan abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Serum ferritin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine albumin/creatinine ratio increased (Investigations) | 2 | 1 | 3 | 1 | 5 | 1 | 1 | 0 | 0 | 0
Urine leukocyte esterase (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3 | 4 | 2 | 1 | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ketosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 6 | 2 | 2 | 2 | 2 | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1 | 7 | 2 | 4 | 3 | 5 | 3 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 2 | 0 | 2 | 1 | 3 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign neoplasm of conjunctiva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 2 | 0 | 3 | 1 | 1 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyposmia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 2 | 3 | 1 | 1 | 1 | 1 | 2 | 2
Binge drinking (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 2
Grief reaction (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Organic brain syndrome (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 0 | 3 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 1 | 2 | 1 | 3 | 0 | 1 | 0 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 3
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast haematoma (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epididymal cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulval disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 0 | 1 | 1 | 2 | 0 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT03100058/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT03100058/SAP_001.pdf